CLINICAL TRIAL: NCT00754104
Title: A Phase 1, Open Label Study of ABT-869 in Combination With Tarceva in Subjects With Advanced Non-hematologic Malignancy
Brief Title: Study of ABT-869 in Combination With Tarceva in Subjects With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Rod Humerickhouse, Global Project Head, Oncology, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-371
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — linifanib; Erlotinib Hydrochloride

ARMS (1):
- A (Experimental)
  Interventions: Drug: ABT-869; Drug: Tarceva

INTERVENTIONS:
Drug: ABT-869 — 0.25 mg/kg. daily.
Drug: Tarceva — 150mg, daily.

SUMMARY:
Study of ABT-869 in Combination with Tarceva in Subjects with Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a histologically or cytologically confirmed non-hematologic malignancy.
* Subject must have an ECOG Score of 0-2.
* Adequate organ function.

Exclusion Criteria:

* Subject has received targeted VEGF/PDGF therapy (tyrosine kinase inhibitor) therapy. Prior Avastin allowed.
* Subject has untreated brain or meningeal metastases.
* History of greater than 10% weight loss.
* Has clinically relevant hemoptysis.
* Subject has proteinuria CTC grade > 1.
* Must not have had radiation therapy or major surgery within 21 days of study day 1.
* The subject currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure (DBP) > 100 mmHg or systolic blood pressure (SBP) > 150 mmHg. Subjects may be re-screened if blood pressure is shown to be controlled with or without intervention.
* The subject has a documented left ventricular ejection fraction (LVEF) < 50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Day 7, 15, 21, 35 and Day 1 of every 8 weeks